CLINICAL TRIAL: NCT07288008
Title: Transcranial Alternating Current Stimulation (tACS) for the Treatment of Anxiety in Veterans: An Open-Label Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham VA Health Care System (U.S. Federal Agency)
Collaborators: Fisher Wallace Laboratories (Industry)
Responsible Party: Principal Investigator, Lori L. Davis, Senior Research Psychiatrist, Birmingham VA Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1893439
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Anxiety; Veterans; Transcranial Alternation Current Stimulation; Post-traumatic stress disorder
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Transcranial Alternating Current Stimulation device (Experimental): Fisher Wallace FW-200 Stimulator, a wearable, battery-powered (2 AA) tACS device comprised of a handheld pulse generator, 2 electrodes that attach to the pulse generator via wires, and an adjustable headband used to secure the electrodes. The tACS device delivers 2 mA (±10% tolerance) of pulsed alternating current, with a pulse width of 33.3 microseconds, using a rectangular, bipolar (bidirectional) waveform, employing a 15,000-Hz carrier frequency and 2 modulating frequencies of 500 Hz and 15 Hz, delivered through two 1.5-inch-diameter (circular) sponge electrodes moistened with tap water and secured under the headband at the squamous temporal bone above the posterior aspect of the zygomatic arch on either side of the head (i.e., center of each electrode located, respectively, at EEG coordinates FTT7h and FTT8h) . The device turns off automatically after each 20-minute treatment session.
  Interventions: Device: Transcranial alternating current stimulator

INTERVENTIONS:
Device: Transcranial alternating current stimulator — Fisher Wallace FW-200 Stimulator, a wearable, battery-powered (2 AA) tACS device comprised of a handheld pulse generator, 2 electrodes that attach to the pulse generator via wires, and an adjustable headband used to secure the electrodes. The tACS device delivers 2 mA (±10% tolerance) of pulsed alternating current, with a pulse width of 33.3 microseconds, using a rectangular, bipolar (bidirectional) waveform, employing a 15,000-Hz carrier frequency and 2 modulating frequencies of 500 Hz and 15 Hz, delivered through two 1.5-inch-diameter (circular) sponge electrodes moistened with tap water and secured under the headband at the squamous temporal bone above the posterior aspect of the zygomatic arch on either side of the head (i.e., center of each electrode located, respectively, at EEG coordinates FTT7h and FTT8h) . The device turns off automatically after each 20-minute treatment session.

SUMMARY:
Transcranial alternating current stimulation (tACS) in a wearable brain stimulation device that delivers a low intensity, pulsed, alternating current via scalp electrodes. Prior sham-controlled clinical trials have shown the therapeutic effects and safety of tACS for the treatment of anxiety and depression. In addition, tACS is rapid acting and well tolerated. After the device is issued to the patient during an in-office orientation and training session, the tACS device can be safely used by the patient at the convenience of their own home. Up to 40 Veterans under that age of 70 who have clinically significant anxiety will be enrolled in an 8-week open-label trial of Model FW-200 tACS to evaluate feasibility, acceptability, adherence and impact on anxiety, depression, post-traumatic stress disorder (PTSD), sleep and neurocognitive measures. Participants may have a concurrent diagnosis of major depressive disorder (MDD) and/or PTSD.

DETAILED DESCRIPTION:
Transcranial alternating current stimulation (tACS) in a wearable brain stimulation device that delivers a low intensity, pulsed, alternating current via scalp electrodes. This device is regulated by the Food and Drug Administration (FDA) within the category of cranial electrotherapy stimulation. Prior sham-controlled clinical trials have shown the therapeutic effects and safety of tACS for the treatment of anxiety and depression. In addition, tACS is rapid acting and well tolerated. After the device is issued to the patient during an in-office orientation and training session, the tACS device can be safely used by the patient at the convenience of their own home. More research in Veteran populations and additional outcomes, such as neurocognitive and post-traumatic stress disorder (PTSD) symptoms, is warranted. Methods: Up to 40 Veterans under that age of 70 who have clinically significant anxiety will be enrolled in an 8-week open-label trial of Model FW-200 tACS to evaluate feasibility, acceptability, adherence and impact on anxiety, depression, PTSD, sleep and neurocognitive measures. Participants may have a concurrent diagnosis of major depressive disorder (MDD) and/or PTSD. They may remain on stable doses of existing antidepressants. After baseline assessment, Veterans meeting eligibility criteria will be trained on the use of the Fisher Wallace FW-200 Stimulator, a wearable, battery-powered (2 AA) tACS device comprised of a handheld pulse generator, 2 electrodes that attach to the pulse generator via wires, and an adjustable headband used to secure the electrodes. The tACS device delivers 2 mA (±10% tolerance) of pulsed alternating current, with a pulse width of 33.3 microseconds, using a rectangular, bipolar (bidirectional) waveform, employing a 15,000-Hz carrier frequency and 2 modulating frequencies of 500 Hz and 15 Hz, delivered through two 1.5-inch-diameter (circular) sponge electrodes moistened with tap water and secured under the headband at the squamous temporal bone above the posterior aspect of the zygomatic arch on either side of the head (i.e., center of each electrode located, respectively, at EEG coordinates FTT7h and FTT8h) . The device turns off automatically after each 20-minute treatment session. Participants will be trained in the use of the tACS and instructed to use it for 20 minutes in the morning and at bedtime (twice daily). Outcomes and self-reported adherence will be measured at 2, 4, 6, and 8 weeks. In addition to anxiety, depression and quality of life outcomes, neurocognitive measures will be collected to investigate a new area of possible improvement in Veterans. Significance: Testing a novel device that has shown preliminary effectiveness and safety in treating anxiety and depression in a Veteran population is important for advancing the care of Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the U.S. military
* English-speaking and provides signed informed consent and HIPAA
* Adults ≤70 years of age
* Past week's GAD-7 of ≥10 which represents at least moderate level of anxiety
* If applicable, antidepressants may be continued if taking the concomitant medication for ≥8 weeks and at stable doses for ≥4 weeks
* Participants of child-bearing potential must have negative pregnancy test at entry and must agree to adhere to a medically acceptable method of birth control

Exclusion Criteria:

* Lifetime bipolar type I, schizophrenia spectrum, or other psychotic disorders based on VA medical records
* Current sedative-hypnotic, stimulant, inhalant and/or opioid use disorder within the past 6 months based on VA medical records and clinical interview
* Diagnosis of moderate to severe alcohol and/or cannabis use disorder within past 6 months based on VA medical records and clinical interview
* History of severe traumatic brain injury (TBI), defined by Ohio State University TBI Identification Method
* Dementia or related progressive neurocognitive disorder as per the medical record
* Use of prohibited medications (see list above) in the prior 2 weeks
* Increased risk of suicide that necessitates inpatient treatment, suicidal ideation/behavior endorsed on 6-item Columbia Suicide Severity Rating Scale screening questionnaire (yes" to question 4 or 5; or yes to # 6 as current), and/or suicidal behavior within past 90 days.
* Treatment with electroconvulsive therapy, vagus nerve stimulation, or transcranial magnetic stimulation within the past 6 months
* Implanted central nervous system devices (e.g. deep brain stimulation)
* Implanted cardiac pacemaker
* Trigeminal neuralgia that is currently symptomatic
* Treatment with evidence-based psychotherapy (EBP) for anxiety, depression or PTSD in the past 14 days. If receiving EBP therapy, he/she should complete EBP prior to entering study. Veterans currently engaged in non-EBP, e.g., supportive counseling or skills group therapies, may continue in these if they have been in this treatment for at least 4 weeks prior to baseline assessments.
* Pregnancy during treatment
* Clinically significant medical/surgical illness that would contraindicate use of tACS, e.g. unstable cardiac condition, those who fear electrical stimulation, presence of skin irritation or abrasions around either electrode site, or who have shrapnel fragments near either electrode site.
* Litigating for disability income for a mental disorder outside the VA compensation and pension process

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7-item (GAD-7) | 8 weeks
  Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report rated on a 4-point Likert scale of frequency ranging from 0=not at all to 3=nearly every day. Total score ranges from 0 to 21. A total score is interpreted as follows: ≤4 minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety. The GAD-7 is sensitive to detecting a change in anxiety severity over the course of treatment.

SECONDARY OUTCOMES:
Patient Health Questionnaire for Depression (PHQ-9) | 8 weeks
  Patient Health Questionnaire for Depression (PHQ-9) is a 9-item self-report rating scale that assesses symptoms of depression with scores ranging from 0 to 27 (higher score = greater severity of symptoms) measured on 4-point Likert scale from 0=not at all to 3=almost all the days.

OTHER OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | 8 weeks
  PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report of post-traumatic stress disorder (PTSD) symptoms; score 0-80; higher=more severe.
Pittsburgh Sleep Quality Index | 8 weeks
  Pittsburgh Sleep Quality Index is a 7-item self-report measure of sleep quality and disruption with scores ranging from 0 to 21 (higher = more severe).
Social Roles and Activities - Short Form (SF8a) | 8 weeks
  Social Roles and Activities - Short Form (SF8a) is an 8-item self-report PROMIS assessing domains of family life, leisure, social relationships, and work. Higher scores represent more ability to participate in social activities and roles.
Work and Social Adjustment Scale (WSAS) | 8 weeks
  Work and Social Adjustment Scale (WSAS) is a 5-item self-report of functional outcomes of daily activities and social roles, scored range 0 to 40 with higher score indicating higher levels of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Davis, MD, Principal Investigator — Birmingham VA Health Care System
Locations (1):
- Birmingham VA, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gehrman PR, Bartky EJ, Travers C, Lapidus K. A Fully Remote Randomized Trial of Transcranial Alternating Current Stimulation for the Acute Treatment of Major Depressive Disorder. J Clin Psychiatry. 2024 Apr 22;85(2):23m15078. doi: 10.4088/JCP.23m15078. PMID 38696220
- [Background] Lee SH, Kim YK. Application of Transcranial Direct and Alternating Current Stimulation (tDCS and tACS) on Major Depressive Disorder. Adv Exp Med Biol. 2024;1456:129-143. doi: 10.1007/978-981-97-4402-2_7. PMID 39261427
- See also: Fisher Wallace web site — https://www.fisherwallace.com/